CLINICAL TRIAL: NCT06177366
Title: Development of a Blood Score for Myelofibrosis Staging in BCR:ABL1 Negative Myeloproliferative Neoplasms Using Bone Marrow Biopsy as a Gold Standard
Brief Title: A New Blood Score for Myelofibrosis Staging
Acronym: FIBROMOELLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231007
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with MPN who need a bone marrow biopsy during the management of the disease
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood samples will be collected at diagnosis, in the same time as BOM is performed

SUMMARY:
BCR:ABL1 negative myeloproliferative neoplasms (MPN) include three entities: polycythemia vera, essential thrombocythemia and primitive myelofibrosis. Myelofibrosis is a life-threatening complication in MPN with several therapeutic options including hematopoietic stem cell transplantation (HSCT) which remains the only curative treatment. Bone marrow biopsy with histological analysis allows myelofibrosis identification and staging. However, it is an invasive procedure that remains painful and provides potential haemorrhagic complications. Development of non-invasive biomarkers for myelofibrosis staging could help to better stratify this disease, better define patients' prognosis and lead to optimal cares.

The main aim of this work is to develop a non-invasive blood score including several biomarkers for myelofibrosis staging in MPN using bone marrow biopsy as a gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of BCR::ABL1 negative MPN according to WHO criteria classification
* Indication for bone marrow biopsy
* Non opposition
* Social security affiliation

Exclusion Criteria:

* Non-contributory biopsy
* AML transformation
* Organ fibrosis (liver, lung, kidney…)
* HSCT
* Chronic inflammatory disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with MPN who need a bone marrow biopsy during the management of the disease
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve | At diagnosis
  Area under the receiver operating characteristic (AUROC) curve of the blood score to discriminate absence or mild fibrosis from advanced fibrosis, using histological analysis as a gold standard.

SECONDARY OUTCOMES:
Number of patients | Up to 2 years
  Number of patients initially classify as essential thrombocythemia and refile with primitive myelofibosis diagnosis.

IPD SHARING:
Plan to Share IPD: Undecided